CLINICAL TRIAL: NCT01825070
Title: The Influence of Tart Montmorency Cherries on Indices of Uric Acid Metabolism
Brief Title: Montmorency Cherry Juice and Uric Acid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Glyn Howatson, Dr, Northumbria University
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: RE10-01-12554; 914 (Other: Northumbria University)
Record Dates: First submitted 2013-03-29; First posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Inflammation
Keywords: Montmorency tart cherries; Inflammation; Uric acid
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low dose (Experimental): Montmorency cherry concentrate, 30 mls
  Interventions: Dietary Supplement: Montmorency cherry concentrate
- higher dose (Experimental): Montmorency cherry concentrate, 60 mls
  Interventions: Dietary Supplement: Montmorency cherry concentrate

INTERVENTIONS:
Dietary Supplement: Montmorency cherry concentrate — Tart Montmorency cherry juice concentrate

SUMMARY:
Cherries have been show to possess the ability to reduce uric acid concentrations and inflammation. Tart Montmorency cherries possess a higher concentration of the plant compounds than other cherries and hence makes the expectation possible that Montmorency cherries will lower uric acid and inflammation.

DETAILED DESCRIPTION:
Plasma and urinary uric acid concentration, plasma phytochemical content and inflammatory biomarkers will be measured in order to elucidate the effects of an acute dose of tart cherry juice on indices related to the condition of gout.

Participants will be required to attend the laboratory at a range of time points over two periods of 96 hours, separated by a 7 day washout period, to provide blood samples. In order to provide a baseline sample, participants will attend the laboratory in the morning following an overnight fast and voiding of any urine. Following this participants will be given 30mls (30 mls provides 323 mg/380 µmol of anthocyanins) of tart cherry juice or placebo, diluted with 60 mls of water to consume within 10 minutes. Participants will be required to consume identical dosages of the supplement immediately prior to evening meals and breakfasts (or same time each morning following blood sampling if non-breakfast eater) over the next 96 hours. Further blood and urine samples will be collected at 1, 2, 3, 5, 8, 24, 26, 48, 50, 72, 74 and 96 hours and will require participants to return to the laboratory at each of these time points. Following the first period of supplementation participants will complete a 7 day washout period in which they will not be required to attend the laboratory. Following the washout period they will repeat the supplementation period consuming the supplement they did not receive during the first period.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy males/females between the ages of 18-40 years

Exclusion Criteria:

* underlying clinical pathology

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in uric acid | 0, 1, 2, 3, 5, 8, 24, 26, 48 hours
  measurement of changes in uric acid over a 48h period

SECONDARY OUTCOMES:
Change in C-reactive protein | 0,1,2,3,5,8,24,26,48 hours
  measurement of changes in c-reative protein over a 48h period

OTHER OUTCOMES:
Change in anthocyanins, polyphenolics and creatinine | 0,1,2,3,5,8,24,26,48 hours
  measurement of changes in anthocyanins, polyphenolics and creatinine over a 48h period

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Howatson, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom